CLINICAL TRIAL: NCT04553419
Title: Antibiotic Treatment Of Staphylococcus Aureus In Stable People With CF (ASAP-CF) Clinical Research Protocol
Brief Title: Antibiotic Treatment Of Staphylococcus Aureus In Stable People With CF
Acronym: ASAP-CF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jonathan Rayment, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H19-00836
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Cephalexin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cephalexin (Experimental): Oral cephalexin (available in capsule or suspension format) dosed at 150 mg/kg/day. Doses will be administered 3 times a day for 2 weeks.
  Interventions: Drug: Cephalexin
- Placebo (Placebo Comparator): The placebo will be available in both capsule and suspension format. Doses will be administered 3 times a day for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cephalexin — Cephalexin capsule: TEVA Cephalexin Cephalexin suspension: LUPIN Cephalexin
  Arms: Cephalexin
Drug: Placebo — Cellulose capsules or suspension
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded study that aims to assess the effect of an oral antibiotic called Cephalexin (150 mg/kg/day) compared to placebo in clinically stable children with cystic fibrosis who have grown a bacteria called MSSA (methicillin-susceptible Staphylococcus aureus) over the course of 2 weeks.

A sensitive technique called MBW (multiple breath washout) will be used to look at how well the participants lungs are functioning during the study and to see if the antibiotic improves function. The primary outcome of the study will be the relative change in the MBW measurement (LCI2.5) between day 0 and day 14 of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF as evidenced by one or more clinical feature consistent with the CF phenotype or positive CF newborn screen AND one or more of the following criteria:

   1. A documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis (QPIT)
   2. A documented genotype with two disease-causing mutations in the CFTR gene
2. Age 3 years and over, up to 17th birthday.
3. Weight ≥ 10.0kg
4. No increase in lower respiratory tract symptoms from baseline for 28 days.
5. At least one episode of MSSA growth on airway culture in the past 24 months OR the past 10 airway cultures, which ever is greater.
6. Successful MBW test occasion at the Screening Visit, per the assessment of the Site MBW Operator.
7. Informed consent by participant or parent/legal guardian with written assent where age-appropriate.

Randomization inclusion at each visit(applied after every Study Visit in the Phase 1)

1. Growth of isolated MSSA on bacterial airway culture from this Study Visit, including cultures collected up to 21 days before this study visit.
2. Acceptable MBW test at this Study Visit, per the assessment of the Site MBW Operator.
3. Participant willing to be randomised.

Exclusion Criteria:

1. Change of any respiratory medications within 28 days of enrollment (i.e. recent increase in pancreatic enzyme dosing, or similar, is not an exclusion).
2. Chronic infection with any of the following: Pseudomonas aeruginosa, Burkholderia cepacia complex, Stenotrophomonas maltophilia or Achromobacter spp, MRSA or any non-tuberculous mycobacteria, where chronic infection is defined as ≥50% positive airway cultures over the previous 12 months or the past 4 airway cultures, which ever is greater (latest culture cannot be positive for Pseudomonas auruginosa).
3. Chronic daily antibiotic use (oral, inhaled or intravenous; including azithromycin or cycling month inhaled antibiotics).
4. Systemic corticosteroid use for any indication within 28 days.
5. Allergic bronchopulmonary aspergillosis (ABPA) requiring corticosteroid therapy within 12 months.
6. Known allergy to cephalexin or other cephalosporins.
7. Previous organ transplantation.
8. Clinical findings that, in the opinion of the Site Investigator, would compromise the safety of the participant or the quality of the study data.
9. Known pregnancy or planning to become pregnant during the study.

Randomisation exclusion(applied after every Study Visit in the Phase 1)

1. Increase in respiratory (upper or lower) symptoms from baseline in the previous 28 days.
2. Diagnosis of a pulmonary exacerbation by the treating physician at the Study Visit.
3. Change of any respiratory medications within 28 days.
4. New diagnosis of allergic bronchopulmonary aspergillosis (ABPA) since previous encounter.
5. New use of chronic daily antibiotics since previous encounter.
6. Clinical findings that, in the opinion of the Site Investigator, would compromise the safety of the participant or the quality of the study data.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The relative change in LCI2.5 between day 0 and day 14 (relative change = [LCI2.5 at day 14-LCI2.5 at day 0]/LCI2.5 at day 0). | 14 days from randomization
  Lung clearance index (LCI) as measured using the multiple breath nitrogen washout (MBW) technique with the Exhlayzer D (Eco Medics, Durnten SUI) device.

SECONDARY OUTCOMES:
Time to next pulmonary exacerbation | up to 12 months
Relative change in percent predicted FEV1 between day 0 and day 14 | 14 days from randomization
Absolute change in FEV1 (mL) between day 0 and day 14 | 14 days from randomization
Relative change in LCI5 between day 0 and day 14. | 14 days from randomization
  Lung clearance index (LCI) as measured using the multiple breath nitrogen washout (MBW) technique with the Exhlayzer D (Eco Medics, Durnten SUI) device.
Absolute change in the CFQ-R(R) between day 0 and day 14. | up to 12 months
  Cystic fibrosis questionnaire - revised (respiratory domain)
MSSA airway culture positivity at day 14 | 14 days from randomization
Time until next growth of MSSA on clinical microbiology samples | up to 12 months
Number of new CF respiratory pathogens (P. aeruginosa etc) from clinical respiratory samples | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rayment, MDCM, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - The Hospital For Sick Children, Toronto, Ontario